CLINICAL TRIAL: NCT04858074
Title: A Proof of Concept (POC) Study to Investigate the Effect of 100% Hypoestes Rosea Powder in Parkinson's Disease Using ActiGraph Wearable as a Quantitative Assessment Tool.
Brief Title: Study to Investigate the Effect of Hypoestes Rosea Powder in Parkinson's Disease
Acronym: PECKO-D
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Ibadan (Other)
Responsible Party: Principal Investigator, ADESOLA OGUNNIYI, Professor, University of Ibadan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UI/EC/20/0320
Record Dates: First submitted 2021-04-07; First posted 2021-04-26 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
Keywords: Motor symptoms; Hoehn and Yahr Stages 1-3; Hypoestes; Sub-Saharan Africa
MeSH Terms: conditions — Parkinson Disease | interventions — hypoestoxide

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled cross-over study
Who Masked: Participant, Investigator
Masking Description: Data recorded by computer application remotely. Investigator will not be aware of patient group; the active and placebo medications are alike
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active medication- PECKO-D (Experimental): Participants will be randomly allocated to experimental drug
  Interventions: Drug: Hypoestoxide
- Placebo (Placebo Comparator): Corn-Starch will be administered as placebo agent
  Interventions: Drug: Hypoestoxide

INTERVENTIONS:
Drug: Hypoestoxide — Its active pharmaceutical ingredient (API) is Hypoestoxide, discovered in 1983, which was recently shown to be active against alpha synuclein and was very effective in modifying disease progression in a transgenic mouse model of PD
  Other Names: PECKO-D forte

SUMMARY:
Parkinson's disease (PD) is a progressive neurological disease characterized by resting tremors, limb stiffness, impaired balance, and slow movement. There is no known cure for PD although levo-3,4 dihydroxyphenylalanine (L-DOPA) and dopamine agonists are effective for improving PD symptoms in the early years following diagnosis. Hypoestes rosea is an evergreen shrub which has anti-inflammatory, anticancer and antimalarial properties. Recent studies showed that the active pharmaceutical ingredient (API) of Hypoestes rosea, Hypoestoxide, was effective in modifying disease progression in a transgenic mouse model of PD.

The aim of this study is to determine the efficacy of Hypoestoxide, as contained in Hypoestes rosea dry leaf powder, in improving motor symptoms in consenting PD patients. The study design is a double-blind, placebo-controlled cross-over trial involving 30 patients with mild to moderate disease (Stages 1-3 of Hoehn and Yahr scale over an 8-week period. The symptoms of the participants will be monitored using mobile phones with an established quantitative assessment tool, mPower2.0, which was previously developed for monitoring symptoms and disease progression in PD patients. In addition, the motor examination component of the International Movement Disorders Society scale will be administered and correlated with the finding on the mobile phone. The outcome measure is an improvement in the motor variables of the study participants with a 10% change from baseline over the 8 weeks of using Hypoestes.

DETAILED DESCRIPTION:
Justification Age-associated disorders are increasing in many low- and middle-income countries due to population ageing and changing lifestyles. PD is a devastating condition which, in the advanced stages, is associated with immobility and uncontrollable tremors. Life then becomes miserable for the sufferers. Unfortunately, there is no cure for the disease except control of symptoms with medications. Any treatment combination that leads to better symptom control will go a long way in improving the quality of life for PD patients. This proof-of-concept study (POC), if successful will give a new lease on life to PD patients. Hence it is considered worthwhile to treat PD patients with a new compound that is contained in a local plant that is readily available and holds promise for efficacy based on its mode of action specifically in reducing the formation of alpha synuclein which underlies the neuronal death in PD.

OBJECTIVES OF THE STUDY

The aim of this study is to determine the efficacy of Hypoestoxide, as contained in Hypoestes rosea dry leaf powder (PECKO-D), in improving motor symptoms in consenting PD patients over an 8-week period.

Specific Objectives:

• To determine the efficacy of Hypoestes rosea in improving motor performance of PD patients through traditional clinical evaluation, use of the selected components of the Motor Examination section of the International Movement Disorders Society Scale and ActiGraph wearable as a quantitative assessment tool.

* To document the side effect profile of the herbal product

Methodology Study site: University College Hospital, Ibadan Study design: Single-center, randomized, double-blind, placebo-controlled trial Study Type: Interventional (Clinical Trial) Allocation: Randomized Masking: Double Primary Purpose: Treatment Study participants: Patients with mild to moderate Parkinson's disease symptoms.

Eligibility Criteria Ages eligible for study: 30 years and older (Adult, older adult) Sexes Eligible for Study: All Accepts healthy volunteers: No Sample size: Being a proof-of-concept study, 19 PD patients will participate in this phase of the study

Inclusion criteria:

• Willing and able to give informed consent.

* Willingness and ability to comply with study requirements.
* PD diagnosis must be confirmed by bradykinesia plus one of the other cardinal signs (resting tremor, rigidity, postural instability) being present.
* Age >30 years
* Men and women with mild to moderate PD: Hoehn and Yahr scale stages 1 - 3. Participants may be on current therapeutic agents (including levodopa, dopamine agonists, anticholinergics, amantadine or selegiline) to treat PD symptoms at the time of enrollment and may remain on these agents throughout the 5-month study period.
* Women of childbearing potential (i.e., those not postmenopausal or surgically sterile) may participate provided that they are using adequate birth control methods for the duration of the study. Women of childbearing potential must have a negative pregnancy test at baseline and be non-lactating.

Exclusion:

* Subjects with advanced, severe disease, including those with dementia, severe osteoarthritis, allergies, stroke, and visual impairment.
* Presence of atypical PD syndromes due to drugs (e.g., metoclopramide, flunarizine), metabolic identified neurogenetic disorders (e.g., Wilson's disease), encephalitis, or other degenerative diseases (e.g., progressive supranuclear palsy).
* Any clinically significant medical condition (e.g., active neoplasm, angina) or laboratory abnormality, which would in the judgement of the investigator interfere with the subjects' ability to participate in the study or be followed.

Study Procedure:

In this study, participants with mild to moderate PD, whether treated or untreated, will be randomized into one of two study arms following an initial baseline assessment to determine motor activity status of each participant as follows:

Baseline Determination: Measurement of motor activities of all participants will be determined for 3 weeks while on regular PD medication(s). The International Movement Disorders Society Scale - Motor Examination (10 selected items on Slowness, Posture, Tremor, Rigidity and Gait) will be utilized for the quantitation of the motor activities.

Drug arm: 15 patients will receive 4 capsules each containing 350 mg orally twice a day of PECKO-D Forte for 8 weeks as add-on therapy to patients' regular PD medication(s).

Placebo arm: 15 participants will receive 4 capsules orally twice a day of United States Pharmacopeia (USP)-grade starch for 8 weeks as add-on to regular PD medication(s).

Wash-Out: Wash-out will be for a duration of 4 weeks in which patients assigned to both arms will take no capsules.

The Switch over: Following the wash-out period, the PECKO-D Forte group will receive 4 capsules of USP-grade starch powder taken orally twice a day for 8 weeks. The placebo group will receive 4 capsules of PECKO-D forte taken orally twice a day for 8 weeks.

Symptoms of the participants will be monitored using traditional clinical evaluation and daily using ActiGraph as an established quantitative assessment tool Once enrolled and given the ActiGraph kit, the participants will be asked to perform four (4) separate study tasks daily during the baseline determination period and throughout the treatment period: gait, tremor, tapping and balance. The International Movement Disorders Society Scale (MDS) - Motor Examination (10 selected items on Slowness, Posture, Tremor, Rigidity and Gait) will be utilized for the quantitation of the motor activities. Data collected using the ActiGraph will be computer-analyzed and the MDS - Motor items will then be analyzed for significant changes in symptom severity relative to baseline status.

Measurements:

These include compliance, gait and balance measures before, during, and after treatment with PECKO-D. Participants will remain on their standard of care PD medications throughout the POC study and possible adverse side effects of the PEKO-D will be monitored.

The following variables will be documented for each of these key measures:

i) Compliance: hours of device worn per day hours of device wear compliance per week hours of device worn per treatment period hours of device worn over the course of the study

ii) Gait measures:

start time of walking period in milliseconds end time of walking period in milliseconds Duration of walking period in seconds Distance walked per walking period in meters Average gait speed per walking period in meters Number of steps per walking period Average stride period per walking period in seconds Freeze index per walking period

iii) Balance measures per detected walking period:

* X (lateral) axis variability in g
* Y (forward) axis variability in g
* Z (vertical) axis variability in g
* X-Y (horizontal) variability in g
* Freeze Index (ratio)

OUTCOME MEASURE: 10% Mean change in motor assessment parameters using the International Movement Disorders Society Scale - selected motor examination items while on the Hypoestes. This equates to 1- to 2-point improvement in motor performance over a 2-month period on Hypoestes in the absence of side effects which will be monitored using pharmacovigilance tools.

Total duration of study: 5 months (2 months on active drugs, 2 months on placebo with one month wash-out period in-between)

The protocol for the study:

PROOF OF CONCEPT STUDY: to investigate the effect of PECKO-D Forte (100% Hypoestes rosea powder) in Parkinson's Disease using ActiGraph GT9X wearable as a quantitative assessment tool

Study Protocol

Serial Number: Hospital Number:

1. Name:
2. Address:
3. Phone number:
4. Gender: Male Female
5. Age (in years) Date of Birth (if known):

   CLINICAL DETAILS:
6. Age at diagnosis of PD:
7. DURATION OF DISEASE AT DIAGNOSIS
8. What are the predominant symptoms? (check all that apply) I) Tremor _______ ii) Stiffness _______iii) Slowness ______iv) Postural instability_______
9. Stage of the disease (from Hoehn and Yahr Scale): _______________ I Unilateral disease only II Bilateral mild disease III Bilateral disease + early impairment of postural stability IV Severe disease requiring considerable assistance V Confinement to wheelchair or bed unless aided
10. Medical co-morbidities i) Hypertension --------- ii) Diabetes Mellitus________ iii) Heart failure_______iv) Chronic lung disease_________ v) Osteoarthritis _______vi) Glaucoma______ VII) Others_________________________
11. Current medications and dosages:

    I) L-Dopa + carbidopa ii) Anticholinesterase iii) DOPA-agonists (specify) iv) Others (specify)
12. Medication Side effects (if any)
13. Any major disability experienced - Yes No IF yes, check whichever is applicable: Cognitive ______ On and off phenomenon_____ Neuropathic pain_________ Dyskinesia____________ others______________

    WILLINGNESS TO PARTICIPATE IN STUDY: Yes No

    PECKO-D Study

    Objective assessment of motor and non-motor- features in PD patients

    The MDS-sponsored Revision of the Unified Parkinson's Disease Rating Scale

1. Posture: Instructions to examiner: Posture is assessed with the patient standing erect after arising from a chair, during walking, and while being tested for postural reflexes. If you notice poor posture, tell the patient to stand up straight and see if the posture improves (see option 2 below). Rate the worst posture seen in these three observation points. Observe for flexion and side-to-side leaning.

0: Normal: No problems.

1. Slight: Not quite erect, but posture could be normal for older person.
2. Mild: Definite flexion, scoliosis or leaning to one side, but patient can correct posture to normal posture when asked to do so.
3. Moderate: Stooped posture, scoliosis or leaning to one side that cannot be corrected volitionally to a normal posture by the patient.
4. Severe: Flexion, scoliosis or leaning with extreme abnormality of posture.

2. Global spontaneity of movement (body bradykinesia) Instructions to examiner: This global rating combines all observations on slowness, hesitancy, and small amplitude and poverty of movement in general, including a reduction of gesturing and of crossing the legs. This assessment is based on the examiner's global impression after observing for spontaneous gestures while sitting, and the nature of arising and walking.

0: Normal: No problems.

1. Slight: Slight global slowness and poverty of spontaneous movements.
2. Mild: Mild global slowness and poverty of spontaneous movements.
3. Moderate: Moderate global slowness and poverty of spontaneous movements.
4. Severe: Severe global slowness and poverty of spontaneous movements.

3. Rigidity: Instructions to examiner: Rigidity is judged on slow passive movement of major joints with the patient in a relaxed position and the examiner manipulating the limbs and neck. First, test without an activation maneuver. Test and rate neck and each limb separately. For arms, test the wrist and elbow joints simultaneously. For legs, test the hip and knee joints simultaneously. If no rigidity is detected, use an activation maneuver such as tapping fingers, fist opening/closing, or heel tapping in a limb not being tested. Explain to the patient to go as limp as possible as you test for rigidity.

0: Normal: No rigidity.

1. Slight: Rigidity only detected with activation maneuver.
2. Mild: Rigidity detected without the activation maneuver, but full range of motion is easily achieved.
3. Moderate: Rigidity detected without the activation maneuver; full range of motion is achieved with effort.
4. Severe: Rigidity detected without the activation maneuver and full range of motion not achieved.

4. Finger tapping: Instructions to examiner: Each hand is tested separately. Demonstrate the task, but do not continue to perform the task while the patient is being tested. Instruct the patient to tap the index finger on the thumb 10 times as quickly AND as big as possible. Rate each side separately, evaluating speed, amplitude, hesitations, halts, and decrementing amplitude.

0: Normal: No problems.

1. Slight: Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the tapping movement; b) slight slowing; c) the amplitude decrements near the end of the 10 taps.
2. Mild: Any of the following: a) 3 to 5 interruptions during tapping; b) mild slowing; c) the amplitude decrements midway in the 10-tap sequence.
3. Moderate: Any of the following: a) more than 5 interruptions during tapping or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing; c) the amplitude decrements starting after the 1st tap.
4. Severe: Cannot or can only barely perform the task because of slowing, interruptions, or decrements.

5. Toe tapping Instructions to examiner: Have the patient sit in a straight-backed chair with arms, both feet on the floor. Test each foot separately. Demonstrate the task, but do not continue to perform the task while the patient is being tested. Instruct the patient to place the heel on the ground in a comfortable position and then tap the toes 10 times as big and as fast as possible. Rate each side separately, evaluating speed, amplitude, hesitations, halts, and decrementing amplitude.

0: Normal: No problems.

1. Slight: Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the tapping movement; b) slight slowing; c) amplitude decrements near the end of the ten taps.
2. Mild: Any of the following: a) 3 to 5 interruptions during the tapping movements; b) mild slowing; c) amplitude decrements midway in the task.
3. Moderate: Any of the following: a) more than 5 interruptions during the tapping movements or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing; c) amplitude decrements after the 1st tap.
4. Severe: Cannot or can only barely perform the task because of slowing, interruptions or decrements.

6. Arising from a chair Instructions to examiner: Have the patient sit in a straight-backed chair with arms, with both feet on the floor and sitting back in the chair (if the patient is not too short). Ask the patient to cross his/her arms across the chest and then to stand up. If the patient is not successful, repeat this attempt up to a maximum of two more times. If still unsuccessful, allow the patient to move forward in the chair to arise with arms folded across the chest. Allow only one attempt in this situation. If unsuccessful, allow the patient to push off using his/her hands on the arms of the chair. Allow a maximum of three trials of pushing off. If still not successful, assist the patient to arise. After the patient stands up, observe the posture.

0: Normal: No problems. Able to arise quickly without hesitation.

1. Slight: Arising is slower than normal; or may need more than one attempt; or may need to move forward in the chair to arise. No need to use the arms of the chair.
2. Mild: Pushes self up from the arms of the chair without difficulty.
3. Moderate: Needs to push off but tends to fall back; or may have to try more than one time using the arms of the chair but can get up without help.
4. Severe: Unable to arise without help.

7. Gait Instructions to examiner: Testing gait is best performed by having the patient walking away from and towards the examiner so that both right and left sides of the body can be easily observed simultaneously. The patient should walk at least 10 meters (30 feet), then turn around and return to the examiner. This item measures multiple behaviors: stride amplitude, stride speed, height of foot lift, heel strike during walking, turning, and arm swing, but not freezing. Observe posture for item 1

0: Normal: No problems.

1. Slight: Independent walking with minor gait impairment.
2. Mild: Independent walking but with substantial gait impairment.
3. Moderate: Requires an assistance device for safe walking (walking stick, walker) but not a person.
4. Severe: Cannot walk at all or only with another person's assistance.

8. Postural Stability Instructions to examiner: The test examines the response to sudden body displacement produced by a quick, forceful pull on the shoulders while the patient is standing erect with eyes open and feet comfortably apart and parallel to each other. Test retropulsion. Stand behind the patient and instruct the patient on what is about to happen. Explain that s/he is allowed to take a step backwards to avoid falling. There should be a solid wall behind the examiner, at least 1-2 meters away to allow for the observation of the number of retropulsive steps. The first pull is an instructional demonstration and is purposely milder and not rated. The second time the shoulders are pulled briskly and forcefully towards the examiner with enough force to displace the center of gravity so that patient MUST take a step backwards. The examiner needs to be ready to catch the patient but must stand sufficiently back so as to allow enough room for the patient to take several steps to recover independently. Do not allow the patient to flex the body abnormally forward in anticipation of the pull. Observe for the number of steps backwards or falling. Up to and including two steps for recovery is considered normal, so abnormal ratings begin with three steps. If the patient fails to understand the test, the examiner can repeat the test so that the rating is based on an assessment that the examiner feels reflects the patient's limitations rather than misunderstanding or lack of preparedness. Observe standing posture.

0: Normal: No problems. Recovers with one or two steps.

1. Slight: 3-5 steps, but subject recovers unaided.
2. Mild: More than 5 steps, but subject recovers unaided.
3. Moderate: Stands safely, but with absence of postural response; falls if not caught by examiner.
4. Severe: Very unstable, tends to lose balance spontaneously or with just a gentle pull on the shoulders.

9. Rest tremor amplitude Instructions to examiner: This and the next item have been placed purposefully at the end of the examination to allow the rater to gather observations on rest tremor that may appear at any time during the exam, including when quietly sitting, during walking, and during activities when some body parts are moving but others are at rest. Score the maximum amplitude that is seen at any time as the final score. Rate only the amplitude and not the persistence or the intermittency of the tremor.

As part of this rating, the patient should sit quietly in a chair with the hands placed on the arms of the chair (not in the lap) and the feet comfortably supported on the floor for 10 seconds with no other directives. Rest tremor is assessed separately for all four limbs and also for the lip/jaw. Rate only the maximum amplitude that is seen at any time as the final rating. Extremity ratings

0: Normal: No tremor.

1. Slight: < 1 cm in maximal amplitude.
2. Mild: ≥ 1 cm but < 3 cm in maximal amplitude.
3. Moderate: ≥ 3 cm but < 10 cm in maximal amplitude.
4. Severe: ≥ 10 cm in maximal amplitude.

10. Constancy of rest tremor Instructions to examiner: This item receives one rating for all rest tremor and focuses on the constancy of rest tremor during the examination period when different body parts are variously at rest. It is rated purposefully at the end of the examination so that several minutes of information can be coalesced into the rating.

0: Normal: No tremor.

1. Slight: Tremor at rest is present ≤ 25% of the entire examination period.
2. Mild: Tremor at rest is present 26-50% of the entire examination period.
3. Moderate: Tremor at rest is present 51-75% of the entire examination period.
4. Severe: Tremor at rest is present > 75% of the entire examination period.

   Total Score: (out of 40)

   Additional measures include:

   Compliance, Gait and Balancing before, during, and after treatment with PECKO-D. Participants will remain on their standard of care PD medications throughout the POC study and possible adverse side effects of the PECKO-D will be monitored.

   The following variables will be documented for each of these key measures:

   i) Compliance: hours of device worn per day hours of device wear compliance per week hours of device worn per treatment period hours of device worn over the course of the study

   ii) Gait measures:

   start time of walking period in milliseconds end time of walking period in milliseconds Duration of walking period in seconds Distance walked per walking period in meters Average gait speed per walking period in meters Number of steps per walking period Average stride period per walking period in seconds Freeze index per walking period

   iii) Balance measures per detected walking period:
   * X (lateral) axis variability in g
   * Y (forward) axis variability in g
   * Z (vertical) axis variability in g
   * X-Y (horizontal) variability in g
   * Freeze Index (ratio)

   Any abnormality on neurological examination?:-----------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------------

   Blood Pressure:

   Pulse:

   Weight:

   Randomization:: A. Active medication: B. Placebo

   Mobile Phone serial number: __________________

   Follow up data:

   I) First review at 8 weeks:

   Date scheduled and time:

   Compliance

   Any reported side effects?: ____________________________________________________

   Any benefits noted subjectively?__________________________________________________

   Other comments: ________________________________________________

   Assess motor performance using the MDS Scale- Record the score_______

   II) 4-week washout period: (No study medications to be administered)

   Any comments________________________________________________

   III) Cross-over for 8 weeks with change of study medications (Placebo to active and vice versa)

   Date scheduled and time:

   Compliance

   Any side effects? ____________________________________________________

   Any benefits noted? __________________________________________________

   Other comments: ________________________________________________

   Assess motor performance using MDS scale: Record the score_______

   Study completed: Yes No (If No, give reasons) _____________________

   Date completed:

   Any comments__________________________________________________________

   Name and signature of investigator_____________________________________

   Date: ----------------------------

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent.

  * Willingness and ability to comply with study requirements.
  * PD diagnosis must be confirmed by bradykinesia plus one of the other cardinal signs (resting tremor, rigidity, postural instability) being present.
  * Age >30 years
  * Men and women with mild to moderate PD: Hoehn and Yahr scale stages 1 - 3. Participants may be on current therapeutic agents (including levodopa, dopamine agonists, anticholinergics, amantadine or selegiline) to treat PD symptoms at the time of enrollment and may remain on these agents throughout the 5-month study period.
  * Women of childbearing potential (i.e., those not postmenopausal or surgically sterile) may participate provided that they are using adequate birth control methods for the duration of the study. Women of childbearing potential must have a negative pregnancy test at baseline and be non-lactating.

Exclusion Criteria:

* • Subjects with advanced, severe disease, including those with dementia, severe osteoarthritis, allergies, stroke, and visual impairment.

  * Presence of atypical PD syndromes due to drugs (e.g., metoclopramide, flunarizine), metabolic identified neurogenetic disorders (e.g., Wilson's disease), encephalitis, or other degenerative diseases (e.g., progressive supranuclear palsy).
  * Any clinically significant medical condition (e.g., active neoplasm, angina) or laboratory abnormality, which would in the judgement of the investigator interfere with the subjects' ability to participate in the study or be followed

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
motor manifestations | eight weeks
  10% Mean change in motor assessment parameters using the International Movement Disorders Society Scale - selected motor examination items while on the Hypoestes. This equates to 1- to 2-point improvement in motor performance over a 2-month period

CONTACTS AND LOCATIONS:
Overall Officials: Adesola Ogunniyi, MD, Principal Investigator — College of Medicine, University of Ibadan, Nigeria
Locations (1):
- College of Medicine, University of Ibadan, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Sociodemographic and clinical details as well as recordings of the ActiGraph app will be made available
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Immediately data analysis is completed and for the next 12 months
Access Criteria: participants, research collaborators, monitoring and evaluation team
URL: http://www.com.ui.edu.ng

REFERENCES:
- [Derived] Olalusi OV, Oguntiloye OO, Makanjuola AI, Yaria JO, Chukwuocha I, Akinyemi RO, Ogunniyi A. Assessing the Efficacy of Peko-D Forte as Add-on Therapy for Parkinson's Disease: A Proof of Concept, Double-Blind, Placebo-Controlled Study. West Afr J Med. 2025 Jan 30;42(1):61-66. PMID 40548419